CLINICAL TRIAL: NCT03073707
Title: The Potential Role of the Household Environment as the Reservoir for Invasive Salmonellosis in Children, Kisangani, DR Congo.
Brief Title: Reservoir of Invasive Salmonellosis in Children, DRC
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: KU Leuven (Other); Université de Kisangani (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1113/16
Record Dates: First submitted 2016-11-16; First posted 2017-03-08 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Salmonella Infections; Infection of Bloodstream
Keywords: Non-Typhoid Salmonella; Invasive blood stream infections; Reservoir; Household environment; Children
MeSH Terms: conditions — Salmonella Infections; Sepsis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Household: Sample collection will be anticipated for 20 cases of NTS infections and household/environment in order to analyze 10 combinations of NTS strains in the index patient and its environment
  Interventions: Behavioral: Sample collection

INTERVENTIONS:
Behavioral: Sample collection — Stool samples will be collected from household members of children diagnosed with NTS infection. In addition stool samples of animals and rats will be collected as well as samples of the water supply of the household.

SUMMARY:
Bloodstream infections caused by non-typhoid Salmonella (NTS) are a major killing disease in Sub-Saharan Africa. Despite the high case fatality rate, the main reservoir -human, zoonotic or environmental- for invasive NTS rests unknown.

The main objective of this study is to assess

1. the household environment (household member, cattle and pets, rats) for intestinal carriage of NTS and
2. the household water supply for presence of NTS .

Households of children with proven NTS invasive infection will be addressed.

DETAILED DESCRIPTION:
This study will be a case-based microbiological assessment of the household environment of index patients presenting with NTS infection. Index patients with laboratory confirmed NTS bloodstream infections will be randomly addressed for the collection of samples from their household (household members, animals (domestic animals and rats) and water supply). The collection of those samples will be done as close as possible to the timing of diagnosis in the index patient.

The sites of blood culture collection are the General Hospitals of Makiso and Kabondo and the Centre Hospitalier Village de Pédiatrie. Blood cultures will be drawn by nursing staff according to the standard procedures of the surveillance study. A total of 1500 blood cultures is expected with a positivity rate of 10% (Falay, 2016). According to previous prevalence data in DR Congo, the expected number of NTS in this sample group will be 50 isolates.

The isolates of Salmonella sp. conserved on TSA agar will be shipped to ITM and the molecular identity of the isolates will be determined and pairs of isolates (index patient-household environment) will be compared for clonal identity, by whole genome sequencing or equivalent technique as appropriate.

A database will be completed that contains the study data. Data that can have a link to the patient identity will be coded.

ELIGIBILITY:
Inclusion Criteria:

* Households where at least one child is diagnosed with NTS bloodstream infection
* Willing to give informed consent

Exclusion Criteria:

* Refusal of participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The criteria for blood collection in patients are standardized according to the surveillance study. This study was approved by the ethics committee of DR Congo on 07th July 2015. The surveillance study will identify children with Salmonella bacteremia, who will be approached for participation in the household study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Environmental presence of NTS in household of index patients | 3 months
  Stool samples of rats,animals and household members as well as samples from household water sources will be collected to assess the presence of Salmonella spp.
Genetic relatedness of environmental/household and index patient results | 3 months
  Assessment of genetic relatedness/clonal identity of Salmonella isolates of index patients, household members and the household environment through whole genome sequencing or equivalent techniques.

SECONDARY OUTCOMES:
Potential demonstration of common source of Salmonella infections in the community by sampling of household environment for NTS, guided by the answers given to questionnaires | 3 months
  Questionnaires will be conducted in different household. The answers to the questions raised will guide the collection of samples (targeted to water, environment and animal species)
Public health knowledge for blood stream infections caused by NTS in DR Congo | 3 months
  As a result of targeted training of household members and the community, knowledge about the prevalence of NTS in the environment will increase, with the aim to avoid blood stream infections caused by NTS
Targeted control prevention measures for blood stream infections caused by NTS in DR Congo by training provided by health personnel | 3 months
  If the results of the study point to a common reservoir of Salmonella NTS in the community, targeted training will be given and control measures explained. The latter will largely depend on the source discovered (e.g. undercooked meat, water source)

CONTACTS AND LOCATIONS:
Overall Officials: Dadi Falay, Pediatrician, Principal Investigator — University of Kisangani
Locations (1):
- University of Kisangani, Faculty of Medicine, Kisangani, Tshopo, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falay D, Kuijpers LM, Phoba MF, De Boeck H, Lunguya O, Vakaniaki E, Bertrand S, Mattheus W, Ceyssens PJ, Vanhoof R, Devlieger H, Van Geet C, Verheyen E, Ngbonda D, Jacobs J. Microbiological, clinical and molecular findings of non-typhoidal Salmonella bloodstream infections associated with malaria, Oriental Province, Democratic Republic of the Congo. BMC Infect Dis. 2016 Jun 10;16:271. doi: 10.1186/s12879-016-1604-1. PMID 27286886